CLINICAL TRIAL: NCT00823056
Title: The Effect of Probiotics on Infections in Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Holbaek Sygehus (Other); Dept. of Microbiology, Slagelse University Hospital, Region Zealand,DK (Unknown); Chr Hansen A/S (Unknown); Ferrosan A/S (Unknown)
Responsible Party: Ms. Mette Louise Gyhrs, MD., Paediatr. Depart., Uni. Hosp. Holbaek, Region Zealand,DK, Uni. of CPH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Version 2
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Diarrhoea; Respiratory Diseases
Keywords: Probiotics; Infections; Children
MeSH Terms: conditions — Diarrhea; Respiratory Tract Diseases; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: probiotics
- 2 (Active Comparator)
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — placebo
  Arms: 1
Dietary Supplement: probiotics — 0,53 ml MCT oil containing BB12 and TH4 in daily dosage in 9 months
  Arms: 2

SUMMARY:
Probiotics has been known as a dietary supplement for a long period. Recent clinical trials indicate that probiotics might have an effect in preventing common infection diseases in children.

The investigators hypothesis is: if young children in the age of 6 month to 15 mdr. has a daily intake of a suspension containing probiotics in a period of 9 months, the incidence of diarrhoea and respiratory diseases can be reduced.

DETAILED DESCRIPTION:
Probiotics has been known as a dietary supplement for a long period. Recent clinical trials indicate that probiotics might have an effect in preventing common infection diseases in children.

Our hypothesis is: if young healthy children in the age of 6 month to 15 mdr. has a daily intake of a suspension containing probiotics( BB12 and TH4) in a period of 9 months, the incidence of diarrhoea and respiratory diseases can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children born in University Hospital Holbaek,Hospital North,Region Zealand, Denmark in the period of Jan. 2009 to Oct. 2010
* Gestational age > 36. weeks

Exclusion Criteria:

* Chronical heart or lung conditions
* Short Bowel Syndrome
* CVC (Central Venous Catheter)

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 454 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
fewer infections | 9 months

SECONDARY OUTCOMES:
growth | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Mette L. Gyhrs, MD., Principal Investigator — ph.d student
Locations (1):
- Paediatr. Depart., University Hospital Holbaek, University of Copenhagen, Holbæk, Region Sjælland, Denmark

REFERENCES:
- [Derived] Nielsen AC, Gyhrs ML, Nielsen LP, Pedersen C, Bottiger B. Gastroenteritis and the novel picornaviruses aichi virus, cosavirus, saffold virus, and salivirus in young children. J Clin Virol. 2013 Jul;57(3):239-42. doi: 10.1016/j.jcv.2013.03.015. Epub 2013 Apr 19. PMID 23602437